CLINICAL TRIAL: NCT04823520
Title: Trichloroacetic Acid (TCA) Combined With Microdermabrasion in Treatment of Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Mohamed, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCA & MDA to treat melasma
Record Dates: First submitted 2021-03-18; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Melasma
Keywords: TCA; Chemical peeling; Microdermabrasion; Trichloroacetic acid; MELASMA; MDA
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: (Group 1): 30 patients MDA will be done to one half of the face then TCA 15% will be applied to the whole face.
  (Group 2): 30 patients will receive MDA to one side of the face , TCA 20% will then be applied to the whole face.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 15% concentration (Active Comparator): 30 patients MDA will be done to one half of the face then TCA 15% will be applied to the whole face.
  Interventions: Drug: TCA
- Group 20 % concentration (Active Comparator): 30 patients will receive MDA to one side of the face , TCA 20% will then be applied to the whole face.
  Interventions: Drug: TCA

INTERVENTIONS:
Drug: TCA — All patients will receive 6 sessions at 2 weeks intervals,the half face which will recieve MDA and TCA,MDA will be done before appling TCA.
  Other Names: MIcrodermabrasion (MDA)

SUMMARY:
1. To detect the efficacy and safety of combined TCA and MDA in treating melasma.
2. To compare the efficacy and safety of using different TCA concentrations (15% & 20%) alone and in combination with MDA in treatment of melasma.

DETAILED DESCRIPTION:
Melasma is a common, acquired hypermelanosis that occurs in sun exposed areas, mostly on the face, occasionally on the neck, and rarely on the forearms.

Melasma is generally a clinical diagnosis consisting of symmetric reticulated hypermelanosis in three predominant facial patterns: Centro facial, malar, and mandibular The major clinical pattern in 50-80% of cases is the Centro facial pattern, which affects the forehead, nose, and upper lip .

The malar pattern is restricted to the malar cheeks on the face, while mandibular melasma is present on the jawline and chin .

A newer pattern termed extra-facial melasma can occur on non-facial body parts, including the neck, sternum, forearms, and upper extremities .

Using the Wood's light examination, melasma can be classified into four major histological types depending upon the depth of pigment deposition:The epidermal type, in which the pigmentation is intensified under Wood's light, is the most common type. The epidermal type is the most responsive to treatment.

Key etiologic factors include a genetic predisposition, solar damage, barrier abnormalities, and unique sensitivities to hormonal changes including pregnancy, oral contraceptives, and hormone replacement therapy.

Melasma is often difficult to treat, and the condition may be refractory. Despite a strong therapeutic demand, the treatment of melasma remains highly challenging with inconsistent results and almost constant relapses. The treatment of melasma should include a multimodality approach that incorporates photoprotective agents, antioxidant treatments, skin lighteners, exfoliants, and resurfacing procedures, as needed. Evidence-based studies suggest that first line therapies for melasma encompass intense photoprotection and topical lightening agents.

Many depigmenting agents and other therapies such as chemical peeling are used for treating melasma, in the form of mono or combined therapy .

The most commonly used peeling agents are alpha-hydroxy-acids, glycolic acid, Jessner solution, salicylic acid, trichloroacetic acid (TCA), pyruvic acid and phenol .

Chemical peelings are used on a wide scale in cosmetic field including melasma treatment. They often provide clinicians with flexibility in tailoring treat- ments according to patient needs and satisfaction Chemical peelings are used on a wide scale in cosmetic field including melasma treatment. They often provide clinicians with flexibility in tailoring treat- ments according to patient needs and satisfaction Chemical peelings are used on a wide scale in cosmetic field including melasma treatment. They often provide clinicians with flexibility in tailoring treat- ments according to patient needs and satisfaction. Chemical peelings are used on a wide scale in cosmetic field including melasma treatment. They often provide clinicians with flexibility in tailoring treat- ments according to patient needs and satisfaction.

Chemical peeling is a promising treatment for numerous pigmentary disorders as melasma. It aims to remove the melanin rather than the inhibition of melanocytes or melanogenesis by causing controlled necrosis and subsequent regeneration of the epidermis, apart from remodeling of collagen and elastic fibers in the dermis .

TCA is widely used peeling agent in treatment of hyperpigmentation especially melasma. It is a keratolytic acid which cause precipitation of proteins and coagulation necrosis of the epidermis that leads to reepithelization with replacement of smoother skin with an even skin tone .It is not expensive, stable, not light-sensitive and does not need to be neutralized .

Microdermabrasion (MDA) is a minimally invasive epidermal resurfacing procedure used to treat uneven skin tone/texture, photo aging, striae, melasma, and scars.Microdermabrasion uses a variable flow of vacuum suction to maintain contact with the skin whilst the crystals (or diamond tips) get to work by smoothing and buffing the skin's surface.The crystals (or diamond tips) cause gentle mechanical abrasion to the skin, which ultimately removes the stratum corneum layer of the epidermis. As part of the wound healing process, new epidermis forms with enhanced cosmoses. The technique is considered safe for all Fitzpatrick skin types and complications are minimal. In addition to the cosmetic benefits of MDA, studies have also shown improved skin permeability and enhanced delivery of transdermal medications dosed on an area of the skin treated with MDA. Microdermabrasion removes the stratum corneum, the outermost layer of the epidermis . MDA has also been shown to affect deeper layers of the epidermis and dermis. MDA causes a re-arrangement of melanosomes in the basal layer of the epidermis, flattening of rete ridges at the dermal-epidermal junction, increased collagen fiber density at the dermal-epidermal junction, and vascular ectasia in the reticular dermis .

ELIGIBILITY:
Inclusion Criteria:

1. Adults of 18 years and above with bilateral melasma
2. Clinical diagnosis of melasma.
3. Mental capacity to give informed consent.

Exclusion Criteria:

1. Pregnant or nursing women
2. Current use of hormonal birth control medication or any hormonal therapy
3. History of laser or dermabrasion to the face within 9 months of study enrollment
4. Patients with poor wound healing, recurrent herpes simplex and current skin infection (facial warts, molluscum contagiosum) and history of hypertropic scar/keloids
5. Photosensitivity.
6. Patients with unrealistic expectations All the included patients will be subjected to detailed history taking,dermatological examination and Wood's light examination to estimate the depth (epidermal, dermal or mixed) of melasma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
"EFFICACY of combined Trichloroacetic acid (15% or 20 %) and microdermabrasion in treating melasma " | 3 months
  To detect the efficacy of combined Trichloroacetic acid (15% or 20 %) and microdermabrasion in treating melasma.
  Clinical photographs: Front, right and left views of face of each patient will be photographed at baseline, every two weeks and one month after the last session with and high resolution digital camera in natural light.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bandyopadhyay D. Topical treatment of melasma. Indian J Dermatol. 2009;54(4):303-9. doi: 10.4103/0019-5154.57602. PMID 20101327
- [Background] Sanchez NP, Pathak MA, Sato S, Fitzpatrick TB, Sanchez JL, Mihm MC Jr. Melasma: a clinical, light microscopic, ultrastructural, and immunofluorescence study. J Am Acad Dermatol. 1981 Jun;4(6):698-710. doi: 10.1016/s0190-9622(81)70071-9. PMID 6787100
- [Background] Guinot C, Cheffai S, Latreille J, Dhaoui MA, Youssef S, Jaber K, Nageotte O, Doss N. Aggravating factors for melasma: a prospective study in 197 Tunisian patients. J Eur Acad Dermatol Venereol. 2010 Sep;24(9):1060-9. doi: 10.1111/j.1468-3083.2010.03592.x. Epub 2010 Feb 25. PMID 20202051
- [Background] Tamega Ade A, Miot LD, Bonfietti C, Gige TC, Marques ME, Miot HA. Clinical patterns and epidemiological characteristics of facial melasma in Brazilian women. J Eur Acad Dermatol Venereol. 2013 Feb;27(2):151-6. doi: 10.1111/j.1468-3083.2011.04430.x. Epub 2012 Jan 3. PMID 22212073
- [Background] Mandry Pagan R, Sanchez JL. Mandibular melasma. P R Health Sci J. 2000 Sep;19(3):231-4. PMID 11076368
- [Background] Ritter CG, Fiss DV, Borges da Costa JA, de Carvalho RR, Bauermann G, Cestari TF. Extra-facial melasma: clinical, histopathological, and immunohistochemical case-control study. J Eur Acad Dermatol Venereol. 2013 Sep;27(9):1088-94. doi: 10.1111/j.1468-3083.2012.04655.x. Epub 2012 Jul 24. PMID 22827850
- [Background] Lapeere H, Boone B, Schepper SD.(2018) : Hypomelanosis and hypermelanosis. In: Wolff K,Goldsmith LA, Katz SI, editors.Dermatology in general medicine. 7th ed. New York: McGraw Hill. p. 635
- [Background] Lebwohl M, Heymann W, Berth-Jones J. Treatment of skin disease: Comprehensive therapeutic strategies. St. Louis, MO: Mosby; 2002.
- [Background] Molinar VE, Taylor SC, Pandya AG. What's new in objective assessment and treatment of facial hyperpigmentation? Dermatol Clin. 2014 Apr;32(2):123-35. doi: 10.1016/j.det.2013.12.008. PMID 24679999
- [Background] Jutley GS, Rajaratnam R, Halpern J, Salim A, Emmett C. Systematic review of randomized controlled trials on interventions for melasma: an abridged Cochrane review. J Am Acad Dermatol. 2014 Feb;70(2):369-73. doi: 10.1016/j.jaad.2013.07.044. PMID 24438951